CLINICAL TRIAL: NCT03270085
Title: Randomized, Double Blinded, Placebo Controlled Trial to Understand Efficacy of Colesevelam in Diarrhea Predominant IBS Patients With Bile Acid Malabsorption
Brief Title: Trial to Understand Efficacy of Colesevelam in Diarrhea Predominant IBS Patients With Bile Acid Malabsorption
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Michael Camilleri, MD, Michael Camilleri, M.D. Professor of Medicine, Pharmacology and Physiology, Atherton and Winifred W. Bean Professor, College of Medicine Consultant, Division of Gastroenterology and Hepatology, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 17-004639; R01DK115950 (NIH); UL1TR000135 (NIH)
Record Dates: First submitted 2017-08-07; First posted 2017-09-01 (Actual); Results first posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-03

CONDITIONS: Chronic Diarrhea; Irritable Bowel Syndrome With Diarrhea; Bile Acid Malabsorption
MeSH Terms: interventions — Colesevelam Hydrochloride

STUDY DESIGN:
Intervention Model Description: This is the third specific aim of a program on IBS-D with increased fecal bile acid excretion.
Who Masked: Participant, Care Provider, Investigator
Masking Description: 30 subjects with irritable bowel syndrome and diarrhea and bile acid malabsorption will be randomized into 15 people per group in 4-week double-blind, parallel-group trial to Colesevelam or placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Colesevelam (Active Comparator): Once randomized, subjects will have baseline testing period, treatment period, and treatment testing period the study drug. This consists of nine visits and will be over a period of five to nine weeks.
  Baseline testing period consists of: transit test, 4 day high fat diet with 48 hour stool collection, blood samples, rectosigmoid biopsies, one week stool diary, and medication pick up.
  Treatment period will have subject take the study drug 1875 mg of medication orally twice daily with lunch and supper for 4-5 weeks.
  The last period, is the treatment testing period. This consists of a full transit & urine permeability test, 4 day high fat diet with 48 hour stool collection, blood samples, one week stool diary collection, and the return of the unused medication.
  Interventions: Drug: Colesevelam
- Placebo (Placebo Comparator): Once randomized, subjects will have a baseline testing period, treatment period and treatment testing period with the placebo. This consists of nine visits and will be over a period of five to nine weeks.
  The last period, is the treatment testing period. This consists of a full transit & urine permeability test, 4 day high fat diet with 48 hour stool collection, blood samples, one week stool diary collection, and the return of the unused placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Colesevelam — Colesevelam (Welchol) is approved by the Food and Drug Administration (FDA) for the treatment of high blood cholesterol levels and to treat type 2 diabetes however, Colesevelam is not approved for the use proposed in this study and is considered investigational.
  Arms: Colesevelam
Other: Placebo — A placebo looks exactly like the study drug, but it contains no active ingredient. This is used to learn if the effects seen in research participants are truly from the study drug.
  Arms: Placebo

SUMMARY:
To compare with a randomized trial (n=15 per treatment group), effects of colesevelam and placebo treatment, on colonic transit, bowel functions, permeability and tight junction expression in rectosigmoid mucosa of IBS-D with Bile Acid Malabsorption.

DETAILED DESCRIPTION:
Compare the effects of Colesevelam versus the placebo on diabetic subjects with chronic diarrhea. In this study, diabetic subjects will get either the Colesevelam or the placebo, not both.

The plan is to have about 30 subjects complete this study at Mayo Clinic.

ELIGIBILITY:
Inclusion Criteria:

* Females and males age 18 -75.
* An IBS diagnosis based on the Rome III criteria for at least 3 months, with onset at least 6 months previously, of recurrent abdominal pain or discomfort.
* Biomarkers serum alpha C4 ≥ 40 ng/mL or FGF19 ≤ 80 pg/mL or fecal bile acid >2000 micromoles/48h

Exclusion Criteria:

* IBS patients with known clinically-relevant inflammation.
* IBS patient with known bleeding diathesis
* History of abdominal surgery

Patients participating will not take any of the following disallowed medications for at least 7 days prior to and during the remainder of the study:

* Any treatment specifically taken for IBS-D, including loperamide, cholestyramine, alosetron
* Drugs with a known pharmacological activity at 5-HT4, 5-HT2b or 5-HT3 receptors
* All narcotics
* Anti-cholinergic agents
* Tramadol
* Oral anticoagulants
* Antimuscarinics
* Peppermint oil
* Systemic antibiotics, as well as antibiotics directed at colonic flora such as rifaximin and metronidazole

Gastrointestinal preparations:

* Anti-nausea agents
* Osmotic laxative agents
* Prokinetic agents
* 5-HT3 antagonists

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vijayvargiya P, Camilleri M, Carlson P, Nair A, Nord SL, Ryks M, Rhoten D, Burton D, Busciglio I, Lueke A, Harmsen WS, Donato LJ. Effects of Colesevelam on Bowel Symptoms, Biomarkers, and Colonic Mucosal Gene Expression in Patients With Bile Acid Diarrhea in a Randomized Trial. Clin Gastroenterol Hepatol. 2020 Dec;18(13):2962-2970.e6. doi: 10.1016/j.cgh.2020.02.027. Epub 2020 Feb 21. PMID 32088296
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Colesevelam: Once randomized, subjects will have baseline testing period, treatment period, and treatment testing period the study drug. This consists of nine visits and will be over a period of five to nine weeks.
  Baseline testing: transit test, 4 day high fat diet with 48 hour stool collection, blood samples, rectosigmoid biopsies, one week stool diary, medication pick up.
  Treatment period: subject takes study drug 1875 mg orally twice daily with lunch and supper for 4-5 weeks.
  Treatment testing period: full transit & urine permeability test, 4 day high fat diet with 48 hour stool collection, blood samples, one week stool diary collection, and the return of the unused medication.
  Colesevelam: Colesevelam (Welchol) is approved by the Food and Drug Administration (FDA) for the treatment of high blood cholesterol levels and to treat type 2 diabetes however, Colesevelam is not approved for the use proposed in this study and is considered investigational.
- Placebo: Once randomized, subjects will have a baseline testing period, treatment period and treatment testing period with the placebo. This consists of nine visits and will be over a period of five to nine weeks.
  Treatment testing period: full transit & urine permeability test, 4 day high fat diet with 48 hour stool collection, blood samples, one week stool diary collection, and the return of the unused placebo.
  Placebo: A placebo looks exactly like the study drug, but it contains no active ingredient. This is used to learn if the effects seen in research participants are truly from the study drug.
Period: Overall Study
Arm/Group | Colesevelam | Placebo
Started | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Colesevelam | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 44 [34 to 52] | 56 [40 to 68] | 50 [34 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 15 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m2] | 33.2 [28.0 to 37.6] | 33.6 [28.2 to 36.4] | 33.4 [28.0 to 36.7]

OUTCOME MEASURES:

1. Primary Outcome: Total Fecal Bile Acid (BA) Excretion
Description: Total fecal BA excretion was measured using High Performance Liquid Chromatography (HPLC)/tandem mass spectrometry (MS) where single stool samples obtained at baseline and end of treatment were prepared by assay by HPLC/MS by methanol extraction and results are presented as micromoles per gram (μmoles/g) of stool.
Time Frame: Treatment day 28
Measure: Median (Inter-Quartile Range); unit: μmoles/g
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 15 | 15
μmoles/g | 10.7 [8.2 to 17.4] | 3.6 [2.6 to 7.2]
Statistical Analysis 1: Comparison: Colesevelam vs Placebo; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Stool Consistency
Description: Stool consistency as reported by the participant via daily bowel diaries. Stool consistency was based on Bristol Stool Form Scale (BSFS) where 1 - hard lumps, 2 - lumpy sausage, 3 - cracked sausage, 4 - smooth sausage, 5 - soft lumps, 6 - mushy, and 7 - watery. Stool consistency was averaged for the 28 day treatment period.
Time Frame: Treatment days 1 through 28
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 15 | 15
units on a scale | 4.6 [3.9 to 5.2] | 4.6 [4.3 to 5.0]
Statistical Analysis 1: Comparison: Colesevelam vs Placebo; Test type: Superiority; p = 0.81, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Number of Stools Per Day
Description: The total number of bowel movements as reported by the participant via daily bowel diaries. The number of bowel movements were averaged for the 28 day treatment period.
Time Frame: Treatment days 1 through 28
Measure: Median (Inter-Quartile Range); unit: number of stools per day
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 15 | 15
number of stools per day | 3.1 [1.6 to 3.8] | 2.2 [1.6 to 2.9]
Statistical Analysis 1: Comparison: Colesevelam vs Placebo; Test type: Superiority; p = 0.91, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each subject from baseline to the end of the study, approximately 10 weeks, for a total study duration of approximately 18 months.
Arm/Group | Colesevelam | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT03270085/Prot_SAP_000.pdf